CLINICAL TRIAL: NCT06989450
Title: Digital Patient Support Program for Self-Efficacy and Medication Adherence Amongst Women on Adjuvant Endocrine Treatment for Breast Cancer: A Randomized Controlled Trial
Brief Title: Digital Patient Support Program for Self-efficacy and Medication Adherence in Women on Adjuvant Endocrine Treatment for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidekick Health (Industry)
Collaborators: Landspitali University Hospital (Other); University of Iceland (Other); Icelandic Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BC-99-IS-002; VSN24-126 (Other: Icelandic National Bioethics Committee)
Record Dates: First submitted 2025-01-20; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Cancer
Keywords: Cancer; Breast Cancer; Medication adherence; self-efficacy; lifestyle change; endocrine treatment; digital health application
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, open-label, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded for group assignment at the primary analysis (at 12 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital intervention group (Experimental): Participants will be instructed to download Sidekick Health app and receive a code to access the digital intervention in addition to standard of care, as is defined for the control arm.
  The digital patient support program empowers self-efficacy as well as positive lifestyle change by gamification, altruistic rewards, and engaging content with relevant tasks or missions to be completed. The Sidekick platform includes a medication center, which constitutes of behavioral change educational material and methods aimed at improving adherence.
  Beyond this, all participants in the interventional arm will also receive standard of care as defined for the control arm.
  Interventions: Device: Sidekick digital patient support program for patients with breast cancer; Other: Standard of care for breast cancer patients
- Standard of care - control group (Active Comparator): The participants in the control arm will receive standard-of-care treatment. Standard of care includes adjuvant breast cancer treatment and any optional cancer rehabilitation that is not delivered through a mobile application.
  Interventions: Other: Standard of care for breast cancer patients

INTERVENTIONS:
Device: Sidekick digital patient support program for patients with breast cancer — A digital health program delivered through an app that provides holistic lifestyle intervention and medication adherence support.
  Arms: Digital intervention group
Other: Standard of care for breast cancer patients — Standard of care includes adjuvant breast cancer treatment and optional cancer rehabilitation

SUMMARY:
This is a randomized, controlled study to assess the effect of Sidekick Health's digital program on self-efficacy and medication adherence in breast cancer patients prescribed adjuvant anti-hormonal treatment. Participants will be treated with the digital program in addition to standard of care (SoC), or SoC only.

DETAILED DESCRIPTION:
Sidekick Health has developed a digital patient support tool delivered via mobile application (app), to support people who have been diagnosed with breast cancer with self-efficacy in managing their symptoms and with medication adherence and holistic lifestyle modification. The Sidekick platform includes a medication center, including behavioral change material and tools aimed at improving adherence.

The study will be a 2-arm, parallel-group, randomized (1:1) controlled trial to evaluate the performance of Sidekick's digital patient support program for patients with breast cancer on patients' self-efficacy and medication adherence in women undergoing adjuvant endocrine treatment. 140 participants will be included, and eligible participants will be randomized to receive the Sidekick digital support program plus standard of care, or standard of care only.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years or older) diagnosed with breast cancer of stage I, II or III from 1st September 2023 or later
* Have been prescribed adjuvant endocrine therapy for breast cancer.
* Understands written and spoken Icelandic or English.
* Owns a smart-phone compatible with the Sidekick app and capable to use it
* Willing to download the Sidekick app on the smart-phone and to comply with the study measures and visits according to the protocol.
* Capable of providing informed consent for participating in the study.

Exclusion Criteria:

* Having other concurrent conditions that in the opinion of the oncologist may compromise patient safety or study objectives.
* Concurrent participation in another clinical study in which the study treatment may confound the evaluation of the investigational program.
* Metastatic breast cancer (stage IV)
* Previous experience with Sidekick breast cancer program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy and health education impact | 12 weeks from baseline
  Difference in change in total score of the Health Education Impact Questionnaire (heiQ) between the intervention and control groups.
  The heiQ has 8 subscales and is composed of in total 42 questions with a Likert scale of 4 options where 1 represents "strongly disagree" to 4 "strongly agree". Scores on the heiQ range from 42 to 168, with a lower score representing a low impact on patient education.

SECONDARY OUTCOMES:
Medication adherence according to MARS-5 questionnaire | 12 weeks from baseline
  Group difference in self-reported adherence according to MARS-5 questionnaire at 12 weeks The MARS-5 questionnaire consists of five questions measuring adherence ranging from "never" (5 points) to "always" (1 points), therefore the score has a range from 5 - 25 points with higher score indicating high medication adherence.
Self-efficacy and health-education impact after 24 weeks and 1 year | 24 weeks and 1 year
  Group differences in self-efficacy measured by eight scales of Health Education Impact Questionnaire (heiQ) at 24 weeks and 1 year.
Medication adherence after 24 weeks and 1 year according to MARS-5 | 24 weeks and 1 year
  Group difference in self-reported adherence according to MARS-5 questionnaire after 24 weeks and 1 year.
Adherence (PDC) to adjuvant endocrine treatment over 1 year | 1 year
  Adherence to adjuvant endocrine breast cancer treatment over 1 year based on percentage of days covered (PDC) from data from the Icelandic Medicine Registry.
  The proportion of days covered (PDC) is used to estimate medication adherence by looking at the proportion of days in which a person has access to the medication, over a given period of interest, in this case 1 year.
Medication persistence | 1, 2, 3 and 5 years
  Compare the difference between groups in the proportion of participants still taking antihormonal therapy after 1, 2, 3 and 5 years, based on data from the Icelandic Medicine Registry.
BMI | 12, 24 weeks and 1 year
  Group difference in Body Mass Index (BMI) calculated from self-reported weight and height at 12, 24 weeks and 1 year.
  BMI = weight (kg) ÷ height2 (meters)
Physical activity from IPAQ-SF | 12, 24 weeks and 1 year
  Group difference in self-reported physical activity according to IPAQ-SF at 12, 24 weeks and 1 year.
Endocrine treatment symptom management | 12, 24 weeks and 1 year
  Group difference in total score of Endocrine Therapy Symptoms from Endocrine Symptoms Questionnaire at 12, 24 weeks and 1 year
  The questionnaire is composed of 11 questions, where 10 are answered on a Likert scale of 4 options where 1 represents "not at all" to 4 "very much", and 1 question with a 2-option yes or no.
Work status questionnaire | 12, 24 weeks and 1 year
  Work status is a categorical variable representing participants' self-reported employment condition at each follow-up time point. This outcome will be used to assess potential group differences over time.
  No validation measurement tool is used, only questions regarding participant status.
  Work full time Work part-time 50-99% Work part-time, <50% Not on the labor market And reason for not being on labor market or working part time Sick leave Disability Pension Unemployed Other
In app PRO on sleep, energy, stress, quality of life | 12 and 24 weeks
  One PRO that asks users to rate the quality of sleep, energy level, stress level and quality of life.
  The longitudinal change of in-app ePRO in the intervention group will be analysed for these parameters:
  * quality of sleep
  * energy levels
  * stress levels
  * quality-of-life thermometer
User satisfaction in intervention group by MAUQ | 12 weeks
  Scores in the mHealth App Usability Questionnaire (MAUQ) of the intervention group.
  The MAUQ is an 18-item questionnaire. It is composed of questions with Likert scales of 7 options where 1 represents "strongly disagree" to 7 "strongly agree". Scores on the MAUQ range from 18 to 126, with a higher score representing a higher usability.
Engagement, retention and overall activity in the digital intervention | 12 and 24 weeks
  Percentage of users that are active in the digital program, finish the program and engage with the content of the Sidekick digital Program

CONTACTS AND LOCATIONS:
Overall Officials: Olof Kristjana Bjarnadottir, MD, PhD, Principal Investigator — Landspitali University Hospital
Locations (1):
- Landspitali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No
Anonymized Individual Participant Data may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.